CLINICAL TRIAL: NCT06789627
Title: Indirect CAD/CAM Removable Partial Denture Frameworks: a Comparative Study
Brief Title: Oral Health Related Quality of Life in Cad Metallic and Poly Ether Ether Ketone (Peek) Partial Denture Frameworks in Mandibular Kennedy Class I Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Mahmoud Mohamed Hegazi, Prinicipal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HendHegazi
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2021-03

CONDITIONS: Partial Edentulism; Oral Health-Related Quality of Life
Keywords: CAD/CAM; Digital metallic RPD; patient centered outcomes; 3D printing; PEEK; OHIP-14

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RPD with metallic framework (Active Comparator): Indirectly CAD/CAM produced Metallic framework
  Interventions: Other: RPD with metallic framework
- RPD with PEEK framework (Experimental): Indirectly CAD/CAM produced PEEK framework
  Interventions: Other: RPD with PEEK framework

INTERVENTIONS:
Other: RPD with PEEK framework — Indirectly CAD/CAM produced PEEK framework
  Arms: RPD with PEEK framework
Other: RPD with metallic framework — Indirectly CAD/CAM produced metallic RPD
  Arms: RPD with metallic framework

SUMMARY:
The aim of this study was to compare CAD Poly ether ether ketone (PEEK) RPD to CAD metallic RPD in treating partial edentulism in terms of Oral health related quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral free end saddles in the mandible (Kennedy class I) with the last standing abutment second premolar
* Opposing dentition is fully intact or restored to be intact
* Adequate inter-arch space of at least 7mm
* Angle's class I maxilla-mandibular relationship
* Patients with no periodontal disease and good oral hygiene
* Cooperative patients showing motivation to follow-up

Exclusion Criteria:

* Periodontal affection of the abutment teeth
* Skeletal mal-relationship
* Unmotivated patients to maintain adequate oral hygiene and to follow up---- ---- Patients with neuro-mascular disorders
* Systemic disease affecting periodontal health like uncontrolled diabetes

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Oral Health Related Quality of Life (OHRQoL) | 2 years
  measured by Oral Health Impact Profile- 14 Minimum score 0 , Maximum score 56 higher scores indicate worse OHRQoL

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Giza Governorate, Egypt